CLINICAL TRIAL: NCT06673914
Title: EFFECTS OF OLEUROPEIN ON BLOOD PARAMETERS AND INFLAMMATORY MARKERS IN ADULTS WITH METABOLIC SYNDROME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Gulen Ecem Kalkan, Researcher, Atlas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EcemMS
Record Dates: First submitted 2024-07-23; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Metabolic Syndrome; Insulin Resistance; Obesity, Abdominal; Obesity
Keywords: metabolic syndrome; oleuropein; medical nutrition therapy
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Obesity, Abdominal; Obesity | interventions — oleuropein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group: Diet Group (Active Comparator): Control Group: Diet Group Among those who applied to the clinic, those who want to follow their diet will be randomized into this group. Patients in this group will be followed by a personalized diet and be followed up by a dietician.
  Interventions: Behavioral: Control Group: Diet Group
- Experimental: Oleuropein and Diet Group (Experimental): Among those who applied to the clinic, those who want to follow their diet will be randomized into this group. Patients in this group will be followed by a personalized diet and will receive 2 capsules which100 grams of standardized oleuropein-containing olive leaf extract.
  Interventions: Behavioral: Control Group: Diet Group; Dietary Supplement: Oleuropein and Diet Group

INTERVENTIONS:
Behavioral: Control Group: Diet Group — Patient in "Diet Group" and "Oleuropein and Diet Group" will be given a personalized diet and be followed up by a dietician.
Dietary Supplement: Oleuropein and Diet Group — Dietary Supplement: Oleuropein (Olive Leaf Extract) Patients in "Oleuropein and Diet Group" will receive 200 mg/day oleuropein supplement and personalized diet followed up by a dietician.
  Arms: Experimental: Oleuropein and Diet Group

SUMMARY:
The aim of this study is to determine the effect of 6 weeks supplementation of oleuropein on individuals diagnosed with metabolic syndrome. The baseline and end biochemical parameters and anthropometric measurements will be compared with control subjects.

DETAILED DESCRIPTION:
This study was conducted to investigate the effect of adding oleuropein to the medical nutrition therapy of individuals with metabolic syndrome on their anthropometric measurements and biochemical parameters.

Sub-objectives of the study;

Determining the presence of inflammation in patiens with metabolic syndrome Determination of the effect of diet and diet combined with oleuropein on both fasting blood glucose, insulin and blood lipid profile.

Determination of both anti-inflammatory and antidiabetic effects of oleuropein. Determination of the effect of diet and diet combined with oleuropein on anthropometric measurements.

The aim of this study is to compare the anthropometric measurements and biomarkers of patients with metabolic syndrome as a result of the medical nutrition therpy with consumption of olive leaf extract (2 times a day) that has been contain 100 mg oleuropein for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who volunteer to participate in the study by signing the voluntary consent form
* Diagnosed with Metabolic Syndrome
* Individuals who did not have any infection at the time the study started
* Not consuming any medication
* Not pregnant or lactating
* Women aged 18-49 who have not entered menopause and men in the same age group
* Willing to consume the given extract
* Not allergic or intolerant to olive leaves
* No history of drug use
* People with a BMI below 40 kg/m2

Exclusion Criteria:

* The patient included in the study leaves the study
* Any health issues that may affect the results of the research during the research.
* Occurrence of the problem and/or infection
* Becoming pregnant during the research
* Being in the experimental group and not consuming extract regularly
* Failure to comply with the regulated medical nutrition treatment
* Failure to participate in routine meetings and failure to complete necessary measurements
* Starting to use any medication or nutritional supplement during the study
* Leaving study voluntarily

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Fasting Blood Glucose (mg/dl) at 6 weeks | 6 weeks
  The fasting blood glucose (mg/dl) at the baseline and 6 weeks later noted from the routinely requested tests in the hospital. These values recorded for all groups.
Change from Baseline in the Insulin (uU/mL) at 6 weeks | 6 weeks
  The fasting blood glucose (mg/dl) at the baseline and 6 weeks later noted from the routinely requested tests in the hospital. These values recorded for all groups.
Change from Baseline in the Triglyceride (TG) (mg/dl), high density lipoprotein (HDL-C) (mg/dl), low density lipoprotein (LDL-C) (mg/dl), Total Cholesterol (mg/dl) at 6 weeks | 6 weeks
  Triglyceride (TG) (mg/dl), high density lipoprotein (HDL-C) (mg/dl), low density lipoprotein (LDL-C) (mg/dl), Total Cholesterol (mg/dl) at the baseline and 6 weeks later noted from the routinely requested tests in the hospital. These values recorded for all groups.
Change from Baseline in the HOMA-IR at 6 weeks | 6 weeks
  The fasting blood glucose (mg/dl) and fasting insulin (mU/L) values of the individuals with metabolic syndrome at the baseline and 6 weeks later noted from the routinely requested tests in the hospital. HOMA-IR calculated with the formula (fasting glucose (mg/dl) x fasting insulin (mU/L)) / 405. These values recorded for all groups.
Change from Baseline in the BMI (kg/m2) | 6 weeks
  The body weight (kg) and height (m) of the individuals with metabolic syndrome were measured at the baseline and again after 6 weeks by the researcher, who noted the values in their files. The height of the patients was measured with a fixed height meter at 0.5 cm intervals, with shoes off.
  For body analysis, an 8-electrode bioelectrical impedance (BIA) device, Inbody 270, which performs segmental analysis, was used. Patients were asked to remove all metal items (rings, earrings, bracelets, watches, phones, etc.), any heavy clothing, shoes, and socks before stepping on the device. The device was set to -1.0 kg to account for the remaining clothes.
  From these measurements, body weight, body fat (kg), body fat percentage (%), body muscle (kg), and body water (kg) values were recorded. Body mass index (BMI) was calculated as weight (kg) divided by height (m) squared.
Change from Baseline in the Anthropometric Measurements | 6 weeks
  The anthropometric measurements of the individuals with metabolic syndrome at the baseline and 6 weeks taken by the researcher and noted in their files. These measurements included waist circumference (cm), hip circumference (cm), mid-upper arm circumference (cm), waist-to-height ratio (cm), and waist-to-hip ratio (cm). Waist circumference was measured using an inflexible tape at the umbilicus level after normal exhalation to the nearest 0.1 cm. Hip circumference was measured from the widest area between the waist and the thigh. The waist-to-hip ratio was calculated using the formula waist (cm)/hip (cm), and the waist-to-height ratio was calculated using the formula waist (cm)/height (cm). Mid-upper arm circumference was measured on the left arm of the patients. Neck circumference was measured with the shoulders in a free position from the point where the thyroid cartilage was most protruding.

CONTACTS AND LOCATIONS:
Overall Officials: Gülen Ecem Kalkan, PhD, Principal Investigator — Atlas University; Müveddet Emel Alphan, Prof, Study Director — Atlas University
Locations (1):
- Atlas University, Istanbul, Kağıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No